CLINICAL TRIAL: NCT01853696
Title: Prospective, Randomized Comparison of Corticosteroid Dosing Regimens Following Endothelial Keratoplasty
Brief Title: Comparison of Corticosteroid Dosing Regimens After Endothelial Keratoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cornea Research Foundation of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013-0424
Record Dates: First submitted 2013-05-08; First posted 2013-05-15 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Fuchs' Dystrophy; Corneal Edema
MeSH Terms: conditions — Corneal dystrophy, Fuchs' endothelial, 1; Corneal Edema | interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Loteprednol (Active Comparator): Loteprednol etabonate 0.5% gel applied topically 4 times daily for 2 months, 3 times daily for 1 month, twice daily for one month and once daily for 7 months
  Interventions: Drug: loteprednol etabonate
- Prednisolone acetate (Active Comparator): Prednisolone acetate 1% ophthalmic solution applied 4 times daily for two months, 3 times daily for one month, twice daily for one month, and once daily for 7 months
  Interventions: Drug: prednisolone acetate 1%

INTERVENTIONS:
Drug: loteprednol etabonate
  Other Names: Lotemax gel
  Arms: Loteprednol
Drug: prednisolone acetate 1%
  Arms: Prednisolone acetate

SUMMARY:
Graft rejection has traditionally been one of the leading causes of cornea transplant failure. To help prevent rejection, corticosteroid eye drops are used for an extended period after transplant surgery. The purpose of this study is to compare the efficacy and side effects of different corticosteroid dosing regimens after endothelial keratoplasty (cornea transplant) surgery.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Male or female patient who had endothelial keratoplasty procedure within the past 1 to 7 weeks
* Patient is able and willing to administer eye drops
* Patient is able to comprehend and has signed the Informed Consent form.
* Patient is likely to complete the one-year course of the study

Exclusion Criteria:

* A history of a previous rejection episode in the study eye
* A patient exhibiting intraocular inflammation
* A patient with a known sensitivity to any of the ingredients in the study medications
* A patient who has a condition (i.e., UNCONTROLLED systemic disease) or is in a situation which in the investigator's opinion may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study
* A patient with abnormal eyelid function.
* A patient that is exhibiting active corneal ulceration, keratitis, or conjunctivitis, or who has a history of herpetic keratitis.
* Presence of any ocular disease that would interfere with the evaluation of the study treatment. However, patients with a history of cystoid macular edema, age-related macular degeneration, controlled glaucoma, corneal neovascularization, and other non-interfering comorbidities may be enrolled.
* A patient with a history of non-compliance with using prescribed medication.
* A patient who is concurrently involved in or participated in another randomized clinical trial within 30 days prior to enrollment in this study.
* Patients who are pregnant or planning to become pregnant within the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Price, Jr., MD, Principal Investigator — Price Vision Group
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Price MO, Feng MT, Scanameo A, Price FW Jr. Loteprednol Etabonate 0.5% Gel Vs. Prednisolone Acetate 1% Solution After Descemet Membrane Endothelial Keratoplasty: Prospective Randomized Trial. Cornea. 2015 Aug;34(8):853-8. doi: 10.1097/ICO.0000000000000475. PMID 26020827

RESULTS

PARTICIPANT FLOW:
Groups:
- Loteprednol: Loteprednol etabonate 0.5% gel applied topically 4 times daily for 2 months, 3 times daily for 1 month, twice daily for one month and once daily for 7 months
  loteprednol etabonate 0.5% gel
- Prednisolone Acetate: Prednisolone acetate 1% ophthalmic solution applied 4 times daily for two months, 3 times daily for one month, twice daily for one month, and once daily for 7 months
  prednisolone acetate 1%
Period: Overall Study
Arm/Group | Loteprednol | Prednisolone Acetate
Started | 84 | 83
Completed | 78 | 78
Not Completed | 6 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Loteprednol: Loteprednol etabonate 0.5% gel applied topically 4 times daily for 2 months, 3 times daily for 1 month, twice daily for one month and once daily for 7 months
  loteprednol etabonate
- Total: Total of all reporting groups
Arm/Group | Loteprednol | Prednisolone Acetate | Total
Number analyzed (Participants) | 84 | 83 | 167
Age, Continuous [Median (Full Range); unit: years] | 69 [22 to 88] | 69 [22 to 89] | 69 [22 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 61 | 117
  Male | 28 | 22 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 84 | 82 | 166
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 84 | 83 | 167

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure
Description: Number of eyes in which the absolute intraocular pressure equaled or exceeded 24 mm Hg OR in which there was a relative increase of at least 10 mm Hg over the baseline preoperative reading.
Time Frame: from 1 to 12 months after transplant
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Loteprednol | Prednisolone Acetate
Number analyzed (Participants) | 84 | 83
Number analyzed (eyes) | 116 | 116
eyes | 11 | 27

2. Secondary Outcome: Immunologic Graft Rejection Episode
Description: Rejection episodes were assessed by slit lamp examination and categorized as definite when an endothelial rejection line was detected in a previously clear graft, probable when inflammation (stromal infiltrate, keratic precipitates, cells in the anterior chamber, or ciliary injection) was detected in a previously clear graft without an endothelial rejection line, and possible if central corneal pachymetry increased by 30 microns or more, even if the cornea was clear and no inflammation was detected by slit lamp examination.
Time Frame: within first year after cornea transplantation
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Loteprednol | Prednisolone Acetate
Number analyzed (Participants) | 84 | 83
Number analyzed (eyes) | 116 | 116
eyes | 0 | 0

ADVERSE EVENTS:
Time Frame: 11 months study duration
Arm/Group | Loteprednol | Prednisolone Acetate
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/83
Other Adverse Events (participants affected / at risk) | 0/84 | 0/83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No